CLINICAL TRIAL: NCT07118800
Title: Randomized Phase III Study Evaluating Two Treatment Strategies for Locally Advanced Rectal Cancer in Patients ≥75 Years Old
Brief Title: Study Evaluating Two Treatment Strategies for Rectal Cancer in Patients ≥75 Years Old
Acronym: NACRE-2
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: UNICANCER (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UC-GIG-2408; 2025-521619-37-00 (EU CTIS Number)
Record Dates: First submitted 2025-08-05; First posted 2025-08-12 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-07

CONDITIONS: Locally Advanced Rectal Adenocarcinoma
Keywords: Locally advanced; Rectum; Resectable; Adenocarcinoma; FOLFOX; Total neoadjuvant treatment; watch and wait; Non operative management; Short Course Radiotherapy
MeSH Terms: conditions — Adenocarcinoma | interventions — Fluorouracil; Oxaliplatin; Leucovorin; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Short Course Radiotherapy (SCRT) (Active Comparator): SCRT 25 Gy in 5 fractions of 5 Gy delivered in one week
  Interventions: Radiation: Short Course Radiotherapy
- Short Course Radiotherapy followed by FOLFOX4s (Experimental): SCRT 25Gy in 5 fractions of 5Gy delivered in one week followed by 6 cycles of FOLFOX4s intravenously: Oxaliplatin 85mg/m² over 2h, folinic acid 400mg/m2 (or L-folinic acid 200 mg/m2) over 2h, Fluorouracil "bolus" 400mg/m², Fluorouracil: 2400mg/m² over 46h, every 14 days for 12 weeks (max: 6 cycles). FOLFOX4s regimen will be started 2-4 weeks after completion of radiotherapy.
  Interventions: Drug: FOLFOX4s; Radiation: Short Course Radiotherapy

INTERVENTIONS:
Drug: FOLFOX4s — 6 cycles of FOLFOX4s intravenously: Oxaliplatin 85mg/m² over 2h, folinic acid 400mg/m2 (or L-folinic acid 200 mg/m2) over 2h, Fluorouracil "bolus" 400mg/m², Fluorouracil: 2400mg/m² over 46h, every 14 days for 12 weeks (max: 6 cycles). FOLFOX4 regimen will be started 2-4 weeks after completion of radiotherapy
  Other Names: Chermotherapy; 5FU + Oxaliplatin + folinic acid
  Arms: Short Course Radiotherapy followed by FOLFOX4s
Radiation: Short Course Radiotherapy — 25Gy in 5 fractions of 5Gy delivered in one week (short-course radiotherapy)
  Other Names: SCRT; Radiotherapy

SUMMARY:
The primary objective of the NACRE-2 trial is to assess whether the addition of chemotherapy after short-course radiotherapy is more effective than short-course radiotherapy alone in elderly patients with locally advanced rectal cancer. Secondary objectives will assess the efficacy and safety profile of the combination, as well as its effect on patients' quality of life.

Patients will be separated into two groups to receive their assigned treatment:

* Group 1: Short-duration radiotherapy according to standard practice lasting one week, followed by chemotherapy with FOLFOX4s consisting of oxaliplatin (85 mg/m²), folinic acid (400 mg/m²) and 5-Fluoro-Uracil (400 mg/m² administered in hospital, followed by 2400 mg/m² administered over 46 hours at home) every two weeks for 3 months
* Group 2: Short-duration radiotherapy according to standard practice, lasting one week To receive treatment, patients must come to the hospital where, at each visit, the medical team will carry out medical examinations, prior to administering treatment, to assess the patient's general state of health and tolerance to treatment.

A radiological assessment of the disease will be carried out 11 weeks after the end of radiotherapy. Patients whose tumors have not shrunk will undergo surgery to remove them and enter the follow-up phase. Patients whose tumors have shrunk will not undergo surgery, and will enter a surveillance phase. At 21 weeks, patients whose tumors are still present will undergo surgery and enter the follow-up phase. Patients whose tumors have disappeared will remain in a surveillance phase.

During the surveillance or follow-up phases, patients will be monitored in hospital every 3 months (if no progression is observed). In the case of surgery, patients will be monitored every 6 months. The maximum duration of treatment is 3 years.

DETAILED DESCRIPTION:
Comparative interventional prospective phase III, multicenter, randomised, open-label trial evaluating management strategies of locally advanced rectal cancer treatment with SCRT+/-FOLFOX4s+/-TME to optimize chemotherapy use and increase organ preservation in patients ≥ 75 years

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed diagnosis of adenocarcinoma of the rectum
2. Age ≥75 years
3. WHO performance status 0-1
4. cT3a-b with maximum diameter > 5 cm, T3c-d or cT4 tumor on pretreatment pelvic MRI
5. General condition considered suitable for radical pelvic surgery and a systemic therapy with FOLFOX,
6. Distal part of the tumor ≤10 cm from the anal margin, the measurement done by pelvic MRI
7. Oncogeriatrician approval
8. Adequate biological function defined by:

   1. Neutrophils ≥ 1500/mm3
   2. Platelets ≥ 100 000/mm3
   3. Hemoglobin ≥ 10g/dL
   4. Total bilirubin ≤ 1,5 x ULN
   5. Alkaline phosphatases ≤ 1,5 x ULN
   6. Creatinine clearance >50mL/mn (MDRD)
9. Men must agree to use adequate contraception methods for the duration of study treatment and for within 6 months after completing treatment
10. Patients must be affiliated to a Social Security System (or equivalent).
11. Patient must have signed a written informed consent prior to any trial specific procedures. When the patient is physically unable to give their written consent, a trusted person of their choice, independent from the investigator or the sponsor, can confirm in writing the patient's consent
12. Patients must be willing and able to comply with the protocol for the duration of the study including scheduled visits, treatment plan, laboratory tests and other study procedures.

Exclusion Criteria:

1. Metastatic disease
2. Other cancer within 3 years prior to rectal cancer diagnosis (except for in situ cancer and basal cell carcinoma of the skin)
3. Non resectable cancer, including extension to prostate or extension to perineal muscles
4. History of pelvic irradiation
5. Contraindication to FOLFOX 4s chemotherapy and/or radiotherapy and/or TME surgery
6. Contraindication to MRI
7. Microsatellite instability (MSI) and/or mismatch repair deficiency (dMMR)
8. Complete or partial Dihydropyrimidine Deshydrogenase (DPD) deficiency (uracilemia ≥ 16 ng/mL)
9. Arterial or venous thrombotic or embolic events such as cerebrovascular accident (including transient ischemic attacks), deep vein thrombosis or pulmonary embolism within 6 months before start of treatment
10. Any other serious concomitant disease or disorder that may interfere with the patient's participation in the study and safety during the study (e.g., severe liver, heart, kidney, lung, metabolic, or psychiatric disorders).
11. Concurrent treatment with other experimental drugs or other anti-cancer therapy, treatment in a clinical trial within 30 days prior to randomization
12. Any psychiatric disorder precluding understanding of information of trial related topics and giving informed consent
13. No prior chemotherapy or surgery for rectal cancer
14. Any serious underlying medical condition (as judged by the investigator) that could impair the ability of the patient to participate in the trial
15. Persons deprived of their liberty or under protective custody or guardianship.
16. Patients unwilling or unable to comply with the medical follow-up required by the trial because of geographic, familial, social, or psychological reasons.

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2025-12-15 (Estimated); Primary Completion 2030-12-15 (Estimated); Study Completion 2032-01-15 (Estimated)

PRIMARY OUTCOMES:
TME-free survival | 2 years
  defined as proportion of patients without TME, or non-salvageable pelvic disease, and without permanent diversion stoma. Patients alive at the time of analysis or lost from follow-up will be censored at the date of the latest news.

SECONDARY OUTCOMES:
Rate of clinical Complete Response | 21 weeks
  Defined as the percentage of CR confirmed by central review after 21 weeks divided by the number of patients.
Overall survival | From randomization to death from any cause, up to 2 years.
  The overall survival is the length of time from randomization that patients enrolled in the study are still alive.
Locoregional failure | Time from randomization to locoregional failure, up to 2 years.
  Defined as either an unresectable rectal primary tumor following protocol neoadjuvant treatment, an R2 resection for the rectal primary tumor, or recurrence in the primary tumor bed after an R0-R1 resection. Tumor regrowth in the rectal wall or in regional lymph nodes after a cCR or near-complete response and a period of Watch & Wait or after local scar excision (for ypT0 and T1 tumor) will not be considered a locoregional failure if followed by an R0-R1 resection.
Disease-free survival | 2 years
  Disease-free survival is defined as the delay between date of inclusion and tumor relapse (local, regional, or distant) or death from any cause, whichever occurs first.
Regrowth Rate | 2 years
  defined as the proportion of patients presenting tumor regrowth during their surveillance in the "watch and wait" strategy or after local scar excision after they achieved clinical complete response.
Metastasis-Free Survival | 2 years
  The metastases-free survival is the length of time during and after the treatment for cancer that a patient is still alive and the cancer has not spread to other parts of the body.
Rate of R0 resection | 3 years
  Defined as the percentage of R0 resection among patients with TME surgery (for patient with surgery only)
Rate of postoperative complications of initial surgery | From initial surgery up to 3 months.
  Define as the percentage of patients having complication using Clavien-Dindo classification after initial surgery divided by the number of patients who undergo initial surgery
Rate of postoperative complications of salvage surgey after initial non operative management (NOM) | From salvage surgery up to 3 months.
  Define as the percentage of patients having complication using Clavien-Dindo classification after salvage surgery after initial NOM divided by the number of patients who undergo salvage surgery
Acute and late toxicity during the study | Throughout study completion, up to 3 years.
  The National Cancer Institute-Common Terminology Criteria for Adverse Events version 5 (NCI-CTCAE v5) is widely accepted in the community of oncology research as the leading rating scale for adverse events. This scale, divided into 5 grades (1 = "mild", 2 = "moderate", 3 = "severe", 4 = "life-threatening", and 5 = "death") determined by the investigator, will make it possible to assess the severity of the disorders.
Bowel function | At inclusion, 3 months post-radiotherapy, 12 months and 24 months post inclusion.
  Defined by LARS score
Quality of life questionnaire - Core 30 (QLQ-C30) | at inclusion, 3 months post-radiotherapy, 12 months and 24 months post inclusion.
  Developed by the EORTC, this self-reported questionnaire assesses the health-related quality of life of cancer patients in clinical trials.
  The questionnaire includes five functional scales (physical, everyday activity, cognitive, emotional, and social), three symptom scales (fatigue, pain, nausea and vomiting), a health/quality of life overall scale, and a number of additional elements assessing common symptoms (including dyspnea, loss of appetite, insomnia, constipation, and diarrhea), as well as, the perceived financial impact of the disease.
  All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level.
Quality of life questionnaire - Elderly cancer patients (QLQ-ELD14) | at inclusion, 3 months post-radiotherapy, 12 months and 24 months post inclusion.
  The EORTC QLQ-ELD14, a validated HRQOL questionnaire for cancer patients aged greater than or equal to70 years, is intended to supplement the QLQ-C30.
  The QLQ-ELD14 contains 14 items incorporating five scales to assess mobility, worries about others, future worries, maintaining purpose, and illness burden. In addition, two single items assess joint stiffness and family support. All items are rated on a four-point Likert-type scale (1 = "not at all", 2 = "a little", 3 = "quite a bit", and 4 = "very much"), and are linearly transformed to a 0-100 scale. High scores indicate poor mobility, good family support, much worry about the future, good maintenance of autonomy and purpose, and high burden of illness.
Geriatric Core Dataset (G-CODE) | at 3 months post radiotherapy, 12 and 24 months post inclusion
  The G-CODE was developed by the DIalog for personALization of management in geriatric OncoloGy (DIALOG) intergroup to assess the general health status of the older patient.
  The G-Code contains 10 tools incorporating seven scales to assess social environment, functional status, mobility, nutritional status, cognitive status, depressive mood, and comorbidities. The total scale range 0-62. High score indicate better condition.

CONTACTS AND LOCATIONS:
Overall Officials: Ludovic EVESQUE, Principal Investigator — Centre Antoine Lacassagne

IPD SHARING:
Plan to Share IPD: No
Individual Participant Data will not be shared at an individual level. Those data will be part of the study database including all enrolled patients.